CLINICAL TRIAL: NCT00041223
Title: Double-Blind, Placebo-Controlled, Randomized Phase II Trial of IH636 Grape Seed Proanthocyanidin Extract (GSPE) in Patients With Adverse Effects of High Dose Breast Radiotherapy
Brief Title: IH636 Grape Seed Extract in Treating Hardening of Breast Tissue in Women Who Have Undergone Radiation Therapy for Early Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000069454; RMNHS-GRAPE-1991; RMNHS-1991; EU-20209
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2002-09

CONDITIONS: Breast Cancer; Radiation Fibrosis
Keywords: radiation fibrosis; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Radiation Fibrosis Syndrome | interventions — Grape Seed Proanthocyanidins

INTERVENTIONS:
Dietary Supplement: IH636 grape seed proanthocyanidin extract

SUMMARY:
RATIONALE: IH636 grape seed extract may lessen hardening of breast tissue caused by radiation therapy and may help patients live more comfortably.

PURPOSE: Randomized phase II trial to study the effectiveness of IH636 grape seed extract in treating hardening of breast tissue in women who have undergone radiation therapy for early breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of IH636 grape seed proanthocyanidin extract for the treatment of radiation-induced fibrosis after high-dose radiotherapy in women with a history of early breast cancer.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to time since prior radiotherapy. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral IH636 grape seed proanthocyanidin extract three times daily for 6 months.
* Arm II: Patients receive an oral placebo three times daily for 6 months. Patients are followed at 6 months.

PROJECTED ACCRUAL: A total of 72 patients (48 for arm I and 24 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of early breast cancer

  * T1-T3, N0-N1, M0
* No evidence of cancer recurrence
* Palpable breast induration due to prior radiotherapy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 2 years since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 3 months since prior dietary supplementation containing IH636 grape seed proanthocyanidin extract over 50 mg per day

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, England, United Kingdom